CLINICAL TRIAL: NCT00935493
Title: Guanfacine Treatment for Prefrontal Cognitive Dysfunction in Elderly Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0805003881; R01-030457-1
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Cognitive Aging
Keywords: guanfacine; aging; cognitive aging; prefrontal cognitive function; executive function; prefrontal cortex
MeSH Terms: interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Guanfacine 0.1 mg po qhs (Experimental)
  Interventions: Drug: Guanfacine
- Guanfacine 0.5 mg po qhs (Experimental)
  Interventions: Drug: Guanfacine
- Placebo po qhs (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine — Guanfacine 0.1 mg po qhs
  Arms: Guanfacine 0.1 mg po qhs
Drug: Guanfacine — Guanfacine 0.5 mg po qhs
  Arms: Guanfacine 0.5 mg po qhs
Drug: Placebo — Placebo po qhs
  Arms: Placebo po qhs

SUMMARY:
This proposal aims to determine whether low does of the alpha-2A-adrenoceptor agonist guanfacine can improve deficits in prefrontally-mediated cognitive functions in healthy elderly subjects.

DETAILED DESCRIPTION:
Primary:

* To determine whether low does of the α2A-adrenoceptor agonist guanfacine can improve deficits in prefrontally-mediated working memory and executive control functions, in healthy elderly subjects. Subjects will be randomly assigned to receive placebo or guanfacine at one of two dose levels: 0.1 mg, or 0.5 mg daily at bedtime in double-blind fashion for twelve weeks.

Secondary:

* To determine whether guanfacine can favorably influence global status and quality of life (QOL) in healthy elderly subjects.
* To determine whether low-dose guanfacine is safe and well-tolerated in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled will be nondemented, male and female individuals who meet the following inclusion criteria:

* 75 years of age or older
* Fluent in English
* Stable medical condition for at least 4 weeks prior to Screening visit
* Stable dose of non-excluded medications for at least 4 weeks prior to Screening visit

Exclusion Criteria:

* Dementia
* Mild Cognitive Impairment (Amnestic MCI)
* Clinically significant neurologic disease
* Clinically significant or unstable medical conditions that would interfere with participation in the trial
* Known hypersensitivity to guanfacine
* History of alcohol or substance abuse or dependence within the past 5 years
* Active major psychiatric disorders, including major depression
* History of mental retardation
* Significant abnormalities on clinical laboratories, ECG, or physical examination
* Impairment of visual or auditory acuity sufficient to interfere with completion of study procedures
* Education level < 6 years

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H van Dyck, MD, Principal Investigator — Yale University
Locations (1):
- Alzheimer's Disease Research Unit, Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- See also: Yale ADRU Website — http://alzheimers.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 154 subjects were screened, of which 135 were eligible. Of the 135 eligible, 12 withdrew consent and therefore 123 were randomized.
Period: Overall Study
Arm/Group | Guanfacine 0.1 mg po Qhs | Guanfacine 0.5 mg po Qhs | Placebo po Qhs
Started | 41 | 41 | 41
Completed | 40 | 39 | 40
Not Completed | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Treatment Discontinued | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population consists of the 123 participants (out of 154) that met eligibility requirements and consented to participate in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Guanfacine 0.1 mg po Qhs | Guanfacine 0.5 mg po Qhs | Placebo po Qhs | Total
Number analyzed (Participants) | 41 | 41 | 41 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.0 (4.0) | 80.1 (4.0) | 80.5 (4.0) | 80.2 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 17 | 54
  Male | 22 | 23 | 24 | 69

OUTCOME MEASURES:

1. Primary Outcome: Mean in the Prefrontal Executive Function Z-score (PEF6_6)
Description: The primary outcome measure (PEF6_Z) is the mean of z-scores for 6 executive function tasks (CANTAB: Spatial Working Memory, Stockings of Cambridge, Intradimensiona/Extradimensional Shift, Paired Associates Learning; Stroop Color Word Score, Trail Making Test - B).
  The score is composed of six component scales coded as z scores that measures cognitive functioning in which higher scores represent better cognitive functioning; therefore, the least squares means listed here represent mean outcome changes from baseline
Time Frame: 12 weeks
Population: 119 of the 123 trial participants had outcome data recorded at 12 weeks follow-up.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Groups:
- Guanfacine 0.1 mg: Guanfacine: Guanfacine 0.1 mg
- Guanfacine 0.5 mg: Guanfacine: Guanfacine 0.5 mg
- Placebo: Placebo: Placebo
Arm/Group | Guanfacine 0.1 mg | Guanfacine 0.5 mg | Placebo
Number analyzed (Participants) | 40 | 39 | 40
Z-score | 0.121 (0.056) | 0.213 (0.056) | 0.270 (0.056)
Statistical Analysis 1: Comparison: Guanfacine 0.1 mg vs Placebo; Test type: Superiority or Other; p = 0.06, Regression, Linear
Statistical Analysis 2: Comparison: Guanfacine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.47, Regression, Linear

2. Secondary Outcome: Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC)
Description: The seven-point scale was collapsed into 3 groups and coded as a three-level ordinal scale of global status, representing ordered levels of worse (including minimally, moderately and markedly worse), unchanged, and improved (including minimally, moderately, and markedly improved) global status.
Time Frame: 12 weeks
Population: 119 of the 123 trial participants had outcome data recorded at 12 weeks of follow-up
Measure: Number; unit: participants
Arm/Group | Guanfacine 0.1 mg | Guanfacine 0.5 mg | Placebo
Number analyzed (Participants) | 40 | 39 | 40
participants
  Worse | 4 | 2 | 3
  No Change | 20 | 22 | 25
  Improved | 16 | 15 | 12
Statistical Analysis 1: Comparison: Guanfacine 0.1 mg vs Placebo; Test type: Superiority or Other; p = 0.67, Regression, Logistic
Statistical Analysis 2: Comparison: Guanfacine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.46, Regression, Logistic

3. Secondary Outcome: Quality of Life (SF-36 MCS)
Description: Quality of Life (QOL) was assessed using the SF-36 (36-Item Short-Form Health Survey; QualityMetric, Lincoln, RI), MCS subscale. The SF-36 is a self-administered general health-related quality of life scale with 36 items. The MCS subscale has been shown to be responsive in psychoactive drug trials. The score range is 0-100.
  Higher scores represent better mental health; therefore, the least squares means listed here represent mean outcome changes from baseline.
Time Frame: 12 weeks
Population: 119 of the 123 trial participants had outcome data recorded at 12 weeks of follow up
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Guanfacine 0.1 mg | Guanfacine 0.5 mg | Placebo
Number analyzed (Participants) | 40 | 39 | 40
units on a scale | -0.618 (0.825) | -0.960 (0.835) | -0.083 (0.829)
Statistical Analysis 1: Comparison: Guanfacine 0.1 mg vs Placebo; Test type: Superiority or Other; p = 0.65, Regression, Linear
Statistical Analysis 2: Comparison: Guanfacine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.46, Regression, Linear

ADVERSE EVENTS:
Arm/Group | Guanfacine 0.1 mg | Guanfacine 0.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/41 | 1/41 | 2/41
Other Adverse Events (participants affected / at risk) | 25/41 | 32/41 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guanfacine 0.1 mg (N=41) | Guanfacine 0.5 mg (N=41) | Placebo (N=41)
Speech impairment/Use of right side (Nervous system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Hyponatremia (Blood and lymphatic system disorders) | 0 | 1 | 0
Non-ST Elevation Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Right Frontal Subarachnoid Hemorrhage (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guanfacine 0.1 mg (N=41) | Guanfacine 0.5 mg (N=41) | Placebo (N=41)
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0
Chest Pain (Cardiac disorders) | 0 | 1 | 1
Hypertension (Cardiac disorders) | 1 | 2 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abrasion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Bee Stings (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Bruising (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hair Loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Insect Bite (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Laceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Poison Ivy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Shingles (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Varicose Veins (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cold Sores (General disorders) | 0 | 1 | 0
Dental Implants (General disorders) | 0 | 1 | 1
Dry Mouth (General disorders) | 3 | 7 | 0
Dry Socket (General disorders) | 0 | 1 | 0
Epistaxis (General disorders) | 0 | 1 | 0
Infection Post Tooth Extraction (Infections and infestations) | 0 | 1 | 0
Otitis Media (Ear and labyrinth disorders) | 0 | 1 | 0
Precancerous Lesion On Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rhinorrhea (General disorders) | 1 | 0 | 1
Sinus Congestion (General disorders) | 1 | 0 | 0
Sinusitis (General disorders) | 0 | 0 | 1
Sleep Apnea (General disorders) | 0 | 1 | 0
Sneezing (General disorders) | 0 | 2 | 0
Sore Throat (General disorders) | 1 | 1 | 0
Throat Swelling (General disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Tooth Abscess (General disorders) | 0 | 0 | 1
Hyponatremia (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal Cramps (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1
Anorexia (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 0
Difficulty Swallowing (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 4
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Irregular Bowl Movements (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Allergies (General disorders) | 0 | 0 | 1
Diaphoresis (General disorders) | 0 | 1 | 0
Fall (General disorders) | 2 | 3 | 1
Fever (General disorders) | 0 | 1 | 0
Night Sweats (General disorders) | 1 | 0 | 0
Difficuluty Urinating (Renal and urinary disorders) | 0 | 1 | 0
Diminished Libido (Reproductive system and breast disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 0 | 2 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Leg Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle Strain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Sciatica (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cognitive Worsening (Nervous system disorders) | 1 | 0 | 0
Fatigue (Nervous system disorders) | 3 | 7 | 3
Headache (Nervous system disorders) | 2 | 2 | 1
Insomnia (Nervous system disorders) | 1 | 2 | 1
Ischemic Stroke (Nervous system disorders) | 2 | 0 | 0
Lightheadedness (Nervous system disorders) | 0 | 4 | 4
Sedation (Nervous system disorders) | 3 | 1 | 1
Subarachnoid Hemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Vertigo (Nervous system disorders) | 1 | 0 | 1
Cataracts (Eye disorders) | 2 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Sty (Eye disorders) | 0 | 1 | 0
Subconjunctival Hemorrhage (Eye disorders) | 1 | 0 | 0
Worsening in Near Vision (Eye disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0
Sadness (Psychiatric disorders) | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 9
Urinary Tract Infection (Renal and urinary disorders) | 1 | 1 | 3
Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes